CLINICAL TRIAL: NCT01550029
Title: Targeted Intervention for Bipolar Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-09-14-02; 1K23DA026517-01A1 (NIH)
Record Dates: First submitted 2011-04-21; First posted 2012-03-09 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Nicotine Dependence; Bipolar Disorder
Keywords: Smoking; Tobacco; Nicotine; Bipolar
MeSH Terms: conditions — Tobacco Use Disorder; Bipolar Disorder; Smoking | interventions — Counseling; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counseling/Mood Management (Experimental): A trained counselor will meet with subjects for approximately 60 minutes each week during the 12-week treatment period to provide support for quitting and to help you develop knowledge and skills that can help you quit. Also, subjects will receive the National Cancer Institute's "Clearing the Air" guide to smoking cessation. Some specific areas of focus for this intervention are managing negative moods without smoking and overcoming other obstacles to quitting.
  Interventions: Behavioral: Counseling/Managing Mood
- Counseling/Healthy Lifestyle (Active Comparator): A trained counselor will meet with subjects for approximately 60 minutes each week during the 12-week treatment period to provide support for quitting smoking and to help develop knowledge and skills for quitting. Also, subjects will receive the National Cancer Institute's "Clearing the Air" guide to smoking cessation. Some specific areas of focus for this intervention are developing a better understanding of reasons for smoking and the consequences of tobacco use and identifying ways to establish a healthier lifestyle.
  Interventions: Behavioral: Counseling/Healthy Lifestyle

INTERVENTIONS:
Behavioral: Counseling/Healthy Lifestyle — A trained counselor will meet with subjects for approximately 60 minutes each week during the 12-week treatment period to provide support for quitting and to help develop knowledge and skills for quitting. Also, the National Cancer Institute's "Clearing the Air" guide to smoking cessation will be given to subjects. Some specific areas of focus for this intervention are developing a better understanding of reasons for smoking and the consequences of tobacco use and identifying ways for establishing a healthier lifestyle.
  Other Names: Behavior therapy
  Arms: Counseling/Healthy Lifestyle
Behavioral: Counseling/Managing Mood — A trained counselor will meet with subjects for approximately 60 minutes each week during the 12-week treatment period to provide support for quitting smoking and to help develop knowledge and skills for quitting. Also, subjects will receive the National Cancer Institute's "Clearing the Air" guide to smoking cessation. Some specific areas of focus for this intervention are managing negative moods without smoking and overcoming other obstacles to quitting.
  Other Names: Behavior Therapy
  Arms: Counseling/Mood Management

SUMMARY:
The purpose of this research is to develop and test a new type of smoking cessation counseling for individuals with bipolar disorder.

DETAILED DESCRIPTION:
All participants will receive the nicotine patch, an FDA-approved smoking cessation medication, in an open-label fashion. In addition to the nicotine patch, participants will be randomized to receive one of the two types of counseling for smoking cessation. Participants will be in the research study for approximately 18 weeks. The total number of study visits is 15.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are motivated to quit smoking
* Male or female
* 18 years of age or older
* Diagnosed with bipolar disorder according to DSM-IV criteria
* Stable on medication with no significant changes in the last 3 months before enrollment.
* Smoking 10 cigarettes/day for the past 90 days

Exclusion Criteria:

* Healthy volunteers
* Patients not meeting the criteria for the diagnosis of Bipolar Disorder according to DSM-IV criteria
* Not being and being treated with medication for the bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Prolonged Abstinence from Smoking | Last four weeks of treatment period
  Confirmed prolonged abstinence from smoking during the last 4 weeks of the treatment period.

SECONDARY OUTCOMES:
Prevalence of Abstinence from Smoking | Last 7 days of treatment period
  Prevalence abstinence will be assessed during the last 7 days of treatment period, 7 days prior to follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jaimee Heffner, MD, Principal Investigator — University of Cincinnati
Locations (1):
- The University of Cincinnati, Cincinnati, Ohio, United States